CLINICAL TRIAL: NCT00422253
Title: Will Reduction in Dietary Advanced Glycation End- Products Reduce Chronic Low Grade Inflammation and Improve Insulin Sensitivity in Overweight and Obese Humans
Brief Title: Dietary Advanced Glycation End-products and Insulin Resistance in Overweight and Obese Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 36/06
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2007-01

CONDITIONS: Type 2 Diabetes; Insulin Resistance; Obesity
Keywords: insulin resistance; insulin secretion; advanced glycation end-products
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: dietary intervention

SUMMARY:
We hypothesize that reduction in dietary advance glycation endproducts (AGE) intake will increase insulin sensitivity and normalise insulin secretion in overweight and obese individuals through reduction of chronic low grade inflammation.

We propose to test this hypothesis by performing euglycemic hypeinsulinemic glucose clamp and intravenous glucose tolerance test before and after low AGE diet and normal Australian diet in a cross-over design. This study will provide information relevant to the development and prevention of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* weight stable overweight and obese (BMI ≥ 25kg/m2) non-diabetic individuals, aged 18-50 years and healthy according to medical history, blood biochemistry and physical examination.

Exclusion Criteria:

* Participants will be excluded if they:

  * are aged <18 years or > 50 years;
  * currently smoke, have high alcohol use; or a positive urine drug screening test;
  * have a history of: diabetes, cardiovascular and hematological disease, respiratory, gastrointestinal, endocrine, renal or central nervous system disease, psychosis or psychiatric disorder, active cancer within last 5 years.
  * are actively seeking to lose weight, or if their weight has changed by more than 10 kilograms in the previous 12 months.
  * have been taking medication within one month prior to commencing the study;
  * have acute inflammation (by history, physical or laboratory examination)
  * are on hormonal contraceptives, or pregnant (by HCG urine pregnancy screening test) or lactating
  * have highly unusual dietary habits or follow vegan diets (because of the difficulty in complying with the assigned diet).
  * have current diabetes (determined by history and/or 75g glucose OGTT)
  * are unable to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2006-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbora de Courten, MD PhD, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Baker Heart Research Insitute, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Pearce K, Hatzinikolas A, Moran L, de Courten MPJ, Forbes J, Scheijen JLJM, Schalkwijk CG, Walker K, de Courten B. Disparity in the micronutrient content of diets high or low in advanced glycation end products (AGEs) does not explain changes in insulin sensitivity. Int J Food Sci Nutr. 2017 Dec;68(8):1021-1026. doi: 10.1080/09637486.2017.1319468. Epub 2017 May 2. PMID 28460575
- [Derived] de Courten B, de Courten MP, Soldatos G, Dougherty SL, Straznicky N, Schlaich M, Sourris KC, Chand V, Scheijen JL, Kingwell BA, Cooper ME, Schalkwijk CG, Walker KZ, Forbes JM. Diet low in advanced glycation end products increases insulin sensitivity in healthy overweight individuals: a double-blind, randomized, crossover trial. Am J Clin Nutr. 2016 Jun;103(6):1426-33. doi: 10.3945/ajcn.115.125427. Epub 2016 Mar 30. PMID 27030534
- [Derived] de Courten B, de Courten MP, Schalkwijk CG, Walker KZ, Forbes J. Dietary Advanced Glycation End Products Consumption as a Direct Modulator of Insulin Sensitivity in Overweight Humans: A Study Protocol for a Double-Blind, Randomized, Two Period Cross-Over Trial. JMIR Res Protoc. 2015 Jul 29;4(3):e93. doi: 10.2196/resprot.4552. PMID 26223897